CLINICAL TRIAL: NCT07179302
Title: Comparative Evaluation of LACI and LV Speckle Tracking for Pre- and Post-TAVI Patient Assessment: Advancing Outcome Precision in Aortic Valve Therapy
Brief Title: Pre- and Post-TAVI Patient Assessment: Advancing Outcome Precision in Aortic Valve Therapy
Status: Completed | Type: Observational
Sponsor: Damanhour University (Other)
Collaborators: medina medical center (Other); Tanta University (Other)
Responsible Party: Principal Investigator, Rehab Werida, Associate Professor, Damanhour University
Other Study IDs: Aortic Valve Therapy
Record Dates: First submitted 2025-09-10; First posted 2025-09-17 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TAVI group: Patients undergoing Transcatheter Aortic Valve Implantation.
  Interventions: Procedure: Transcatheter Aortic Valve Implantation (TAVI)

INTERVENTIONS:
Procedure: Transcatheter Aortic Valve Implantation (TAVI) — evaluate the role of the left atrial coupling index (LACI) and left ventricular speckle tracking echocardiography (LVSTE) in enhancing outcome prediction in patients undergoing TAVI.
  Other Names: TAVI

SUMMARY:
The aim of this study is to evaluate the combined utility of the left atrial coupling index (LACI) and left ventricular speckle tracking echocardiography (LVSTE) in improving risk stratification and outcome prediction for patients undergoing Transcatheter Aortic Valve Implantation (TAVI). This study seeks to identify novel prognostic markers that enhance the prediction of mortality, heart failure, and functional recovery, ultimately enabling more personalized clinical decision-making and optimized patient outcomes by integrating the advanced echocardiographic parameters into pre-procedural assessments,.

DETAILED DESCRIPTION:
Transcatheter Aortic Valve Implantation (TAVI) has emerged as a transformative procedure for patients with severe aortic stenosis, particularly those at high surgical risk. However, accurately predicting patient outcomes remains a significant challenge, necessitating improved risk stratification tools. This study aims to evaluate the role of the left atrial coupling index (LACI) and left ventricular speckle tracking echocardiography (LVSTE) in enhancing outcome prediction in patients undergoing TAVI.

By integrating advanced echocardiographic parameters, such as LACI, which reflects left atrial function and ventricular-atrial interaction, and LVSTE, a sensitive measure of myocardial deformation, this research seeks to uncover novel prognostic markers. A prospective cohort of TAVI patients will be studied to assess the association between these indices and post-procedural outcomes, including Repeated hospitalization, heart failure, stroke and myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with severe aortic stenosis and scheduled for TAVI.

Exclusion Criteria:

* Patients with significant mitral or tricuspid valve disease requiring intervention.
* History of atrial fibrillation or other arrhythmias that preclude accurate LACI measurement.
* Poor echocardiographic window preventing reliable imaging.

Ages: 50 Years to 102 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with severe aortic stenosis and scheduled for TAVI will be recruited from Madina Cardiac Center over a period of 12 months Data Collection
  * Baseline Clinical Data: Demographic information, comorbidities, and clinical risk scores
  * Echocardiographic Assessment:
  Pre procedural transthoracic echocardiography (TTE) will be performed to measure: Left Atrial Coupling Index (LACI):
  Left Ventricular Speckle Tracking Echocardiography (LVSTE): Global longitudinal strain (GLS) will be measured to quantify myocardial deformation.
  All echocardiographic measurements will be performed by experienced operators blinded to clinical outcomes.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
Repeated hospitalization in one year | one year
  number of patients need rehospitalization
Need for permanent pacemaker | 6 months
  number of patients need for permanent pacemaker
Myocardial infarction within one year | one year
  incidence of MI in patients
Stroke in one year | one year
  incidence of stroke in patients

CONTACTS AND LOCATIONS:
Overall Officials: Eman Elshaikh, Ass Prof., Study Chair — Madina Cardiac Center, KSA
Locations (2):
- Tanta University, Tanta, Gharbia Governorate, Egypt
- Medina Medical Center, Madinah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu HW, Fortuni F, Butcher SC, van der Kley F, de Weger A, Delgado V, Jukema JW, Bax JJ, Ajmone Marsan N. Prognostic value of left ventricular myocardial work indices in patients with severe aortic stenosis undergoing transcatheter aortic valve replacement. Eur Heart J Cardiovasc Imaging. 2023 Nov 23;24(12):1682-1689. doi: 10.1093/ehjci/jead157. PMID 37409583
- [Background] Takeuchi K, Yamauchi Y, Shiraki H, Sumimoto K, Shono A, Suzuki M, Yamashita K, Toba T, Kawamori H, Otake H, Hirata KI, Tanaka H. Association of acute improvement in left ventricular longitudinal function after transcatheter aortic valve implantation with outcomes for severe aortic stenosis and preserved ejection fraction. J Cardiol. 2023 Oct;82(4):234-239. doi: 10.1016/j.jjcc.2023.04.008. Epub 2023 Apr 19. PMID 37085029